CLINICAL TRIAL: NCT05083806
Title: Multispectral Optoacoustic Tomography for Translational Molecular Imaging in Pompe Disease
Brief Title: MSOT in Pompe Disease
Acronym: SPOT_PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, Study director, University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-238_1-B
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pompe Disease; Pompe Disease (Late-onset); Pompe's Disease Juvenile Onset; Pompe Disease Infantile-Onset
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pompe disease (Experimental): Actual condition
  Interventions: Device: Multispectral Optoacoustic Tomography
- Healthy volunteer (Active Comparator): Healthy control
  Interventions: Device: Multispectral Optoacoustic Tomography

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography — Non-invasive optoacoustic imaging of muscular structure
  Other Names: MSOT; MSOT Echo; MSOT Echo CE

SUMMARY:
In patients with Pompe disease (PD) a progressive abnormal lysosomal glycogen storage in muscle tissue leads to impaired muscle function and to degeneration of muscle fibers. Children and adults with PD present with limb-girdle muscular weakness, diaphragm weakness and impaired breathing ability. Further, patients with classic infantile PD suffer from hypertrophic cardiomyopathy. To date, the muscle pathology and the extent of the disease can be assessed using invasive techniques (e.g., muscle biopsies) or imaging (e.g., MRI). These techniques are time consuming, and especially in young patients, require anesthesia, which increases the acute risk of respiratory failure.

Multispectral optoacoustic tomography (MSOT) allows the detection of specific endogenous chromophores like collagen, myoglobin or hemoglobin by using a non-invasive approach comparable to conventional ultrasound. Instead of sound waves, MSOT illuminates tissue with near-infrared light of transient energy, which is absorbed and results in thermo-elastic expansion of certain molecules. This expansion generates ultrasound waves that are detected by the same device. Multispectral illumination and unmixing then allows the precise localisation and quantification of muscle-specific subcellular structures. MSOT has already been demonstrated the potential to visualize the muscular structure and the clinical extent of muscular disease in patients with Duchenne muscle dystrophy and differentiates those patients from healthy volunteers.

The aim of the study is to establish glycogen as a novel PD-specific imaging target using MSOT-imaging. It intends to identify a PD-specific muscle pathology-signature by quantification of already established targets (collagen, myoglobin, hemoglobin, glycogen if applicable). This signature will aid in differentiating PD from other muscular pathologies and healthy volunteers and will ultimately serve as a potential non-invasive monitoring biomarker.

DETAILED DESCRIPTION:
Pompe disease (PD) is a rare, autosomal-recessive disorder caused by deficiency of the lysosomal acid alpha-glucosidase enzyme (GAA), leading to generalized build-up of glycogen, especially in the heart, muscle, liver and nervous system. Among the glycogen storage diseases, PD is the only one with a defect in lysosomal metabolism.

PD is considered as a progressive disease with variation by age of onset, severity of organ involvement and degree of myopathy. This great phenotypic variability has led to the creation of types based on the age of onset and degree of organ involvement. They all have in common, that symptoms of affected patients are expected to worsen over time if left untreated. The classification is generally based on the age of onset as infantile (infantile onset Pompe disease, IOPD) when it presents during the first 12 months of life and late-onset (LOPD) when first symptoms appear after 12 months of age. If cardiomyopathy is present, IODP is generally referred to as classic Pompe disease (however there may be variably classification in the literature with the infantile or childhood forms). Clinically, infants with classic PD present during the first few months of life with rapidly progressive disease characterized by prominent hypertrophic cardiomyopathy, hepatomegaly, hypotonia, generalized muscle weakness, macroglossia, feeding difficulties and respiratory insufficiency. Mortality rate is high by one year of age if untreated. Patients with non-classic PD will usually present within the first year of life with motor developmental delay and weakness, but without clinically relevant cardiac involvement. The rate of clinical progression is slower in these children and without treatment, death will usually occur in childhood as a result of respiratory insufficiency. LODP include childhood and adult-onset PD. These patients generally present with slowly progressive limb girdle type weakness and respiratory insufficiency without significant cardiomyopathy. The diagnosis of PD is usually established by the typical clinical presentation, followed by confirmation of GAA deficiency in dried blood spots, e.g. through new-born screening. Further (confirmatory) methods include GAA activity measurement in lymphocytes, muscle or skin fibroblasts, as well as GAA mutation testing. All of them are invasive techniques. Early identification is important as it will likely significantly improve the outcome for all patients with PD as treatment can be initiated earlier. Treating the underlying cause of PD involves the replacement of the missing enzyme GAA via enzyme replacement therapy (ERT) with alglucosidase alfa (recombinant human GAA, rhGAA). Currently, this is the only specific treatment approved for PD. In classical IOPD, treatment significantly lengthens survival and improves motor development and respiratory and cardiac function. The sooner ERT begins, the better are the results. With ERT being one very important aspect of care, patients will also need a multidisciplinary approach to ensure that all aspects of the disease are addressed.Regardless of age of onset and severity, all patients with PD should be monitored prospectively. However, there is lack of standardization across centers. A variety of clinical evaluations and tests are currently used for monitoring Pompe's disease, which may include laboratory tests including CK, AST, ALT, and LDH, cardiologic tests including electrocardiogram and echocardiogram and respiratory tests including sleep studies and breathing tests to measure lung capacity. To quantify muscle involvement electromyography is an option as well as clinical tests including 6 minutes walking test or timed to up and go test. Muscle MRI of affected patients often show fatty degeneration of muscles. One study showed that muscle MRI correlates with muscle function in patients with adult-onset Pompe disease. Another study suggested that muscle imaging data in late-onset Pompe disease reveal a correlation between the pre-existing degree of lipomatous muscle alterations and the efficacy of long-term enzyme replacement therapy. For small children, however, there is always a need for sedation for MRI's, limiting its use. Therefore, ultrasound is another option to examine children's muscles.

At the moment there are no prospective biomarkers available to detect muscle degeneration at an early age and/or to follow up disease progression or ERT-treated patients. Within the last years our multidisciplinary research team (Medical Department 1, Department of Pediatrics and Adolescent Medicine, University Hospital Erlangen) published a novel non-invasive imaging modality to be able to detect subcellular tissue composition in vivo. Multi-spectral optoacoustic tomography (MSOT), an imaging technology comparable to ultrasound, allows quantitative imaging in patients of all ages (including the non-sedated child).

ELIGIBILITY:
Inclusion Criteria:

Pompe disease:

* Confirmed diagnosis of Pompe disease
* From 18 years of Age
* Independent from current therapy

Muscular dystrophy:

* Genetically confirmed diagnosis
* From 18 years of Age
* Independent from current therapy

Health volunteer:

* From 18 years of Age, matched (age, gender) to PD collective

Exclusion Criteria:

Pompe disease:

* Pregnancy
* Tattoo on skin to be examined

Muscular dystrophy:

* Pregnancy
* Tattoo on skin to be examined

Health volunteer:

* Anamnestic of other signs of myopathy or liver disease
* Pregnancy
* Tattoo on skin to be examined

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Optoacoustic Absorption Spectrum of Muscle and liver in PD | 60 minutes for MSOT, 1 Visit
  Difference in optoacoustic spectrum in patients compared to healthy volunteers

SECONDARY OUTCOMES:
Quantitative glycogen signal (in arbitrary units) | 60 minutes for MSOT, 1 Visit
  Difference of quantitative glycogen signal in Pompe disease patients compared to muscular dystrophy and healthy control
Quantitative lipid signal (in arbitrary units) | 60 minutes for MSOT, 1 Visit
  Difference of quantitative lipid signal in Pompe disease patients compared to muscular dystrophy and healthy control
Quantitative collagen signal (in arbitrary units) | 60 minutes for MSOT, 1 Visit
  Difference of collagen lipid signal in Pompe disease patients compared to muscular dystrophy and healthy control
Quantitative hemo/myoglobin signal (in arbitrary units) | 60 minutes for MSOT, 1 Visit
  Difference of hemo/myoglobin lipid signal in Pompe disease patients compared to muscular dystrophy and healthy control
Muscle oxygenation (in %) | 60 minutes for MSOT, 1 Visit
  Difference of muscle oxygenation in Pompe disease patients compared to muscular dystrophy and healthy control
Heckmatt scale | 30 minutes for B-mode-ultrasound, 1 Visit
  Difference of Heckmatt scale in Pompe disease patients compared to muscular dystrophy and healthy control
Echogenitiy | 30 minutes for B-mode-ultrasound, 1 Visit
  Difference of Echogenitiy in Pompe disease patients compared to muscular dystrophy and healthy control
Gray Scale Level | 30 minutes for B-mode-ultrasound, 1 Visit
  Difference of Gray Scale Level in Pompe disease patients compared to muscular dystrophy and healthy control
Ultrasound Guided Attenuation Parameter (UGAP) of liver | 30 minutes for B-mode-ultrasound, 1 Visit
  Difference of UGAP in Pompe disease patients compared to muscular dystrophy and healthy control
R-PaAt scale | 10 minutes, 1 Visit
  Difference of R-PaAt scale in Pompe disease patients compared to muscular dystrophy and healthy control
Revised Upper Limb Module (RULM) | 1 hour for total muscle testing, 1 Visit
  Correlation of glycogen detected by MSOT with clinical scores
MRC Muscle Strength Grades | 1 hour for total muscle testing, 1 Visit
  Correlation of glycogen detected by MSOT with clinical scores
6-minute-walk-test | 1 hour for total muscle testing, 1 Visit
  Correlation of glycogen detected by MSOT with clinical scores
Stand-up and go test | 1 hour for total muscle testing, 1 Visit
  Correlation of glycogen detected by MSOT with clinical scores
Quick motor function test | 1 hour for total muscle testing, 1 Visit
  Correlation of glycogen detected by MSOT with clinical scores
Respiratory function test (FEV1, FVC) | 20 minutes, 1 Visit
  Correlation of glycogen detected by MSOT with respiratory function test
Functional. magnetic resonance imaging of lung (Ventilation defect, perfusion defect, combined defects) | 1 hour for total MR Imaging, 1 Visit
  Correlation of glycogen detected by MSOT with functional magnetic resonance imaging parameters
Magnetic resonance imaging of biceps muscle | 1 hour for total MR Imaging, 1 Visit
  Correlation of glycogen detected by MSOT with magnetic resonance imaging parameters

CONTACTS AND LOCATIONS:
Overall Officials: Regina Trollmann, MD, Study Director — University Hospital Erlangen; Ferdinand Knieling, MD, Study Director — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] HERS HG. alpha-Glucosidase deficiency in generalized glycogenstorage disease (Pompe's disease). Biochem J. 1963 Jan;86(1):11-6. doi: 10.1042/bj0860011. No abstract available. PMID 13954110
- [Background] Cupler EJ, Berger KI, Leshner RT, Wolfe GI, Han JJ, Barohn RJ, Kissel JT; AANEM Consensus Committee on Late-onset Pompe Disease. Consensus treatment recommendations for late-onset Pompe disease. Muscle Nerve. 2012 Mar;45(3):319-33. doi: 10.1002/mus.22329. Epub 2011 Dec 15. PMID 22173792
- [Background] Kishnani PS, Steiner RD, Bali D, Berger K, Byrne BJ, Case LE, Crowley JF, Downs S, Howell RR, Kravitz RM, Mackey J, Marsden D, Martins AM, Millington DS, Nicolino M, O'Grady G, Patterson MC, Rapoport DM, Slonim A, Spencer CT, Tifft CJ, Watson MS. Pompe disease diagnosis and management guideline. Genet Med. 2006 May;8(5):267-88. doi: 10.1097/01.gim.0000218152.87434.f3. No abstract available. PMID 16702877
- [Background] Knieling F, Neufert C, Hartmann A, Claussen J, Urich A, Egger C, Vetter M, Fischer S, Pfeifer L, Hagel A, Kielisch C, Gortz RS, Wildner D, Engel M, Rother J, Uter W, Siebler J, Atreya R, Rascher W, Strobel D, Neurath MF, Waldner MJ. Multispectral Optoacoustic Tomography for Assessment of Crohn's Disease Activity. N Engl J Med. 2017 Mar 30;376(13):1292-1294. doi: 10.1056/NEJMc1612455. No abstract available. PMID 28355498
- [Background] Regensburger AP, Fonteyne LM, Jungert J, Wagner AL, Gerhalter T, Nagel AM, Heiss R, Flenkenthaler F, Qurashi M, Neurath MF, Klymiuk N, Kemter E, Frohlich T, Uder M, Woelfle J, Rascher W, Trollmann R, Wolf E, Waldner MJ, Knieling F. Detection of collagens by multispectral optoacoustic tomography as an imaging biomarker for Duchenne muscular dystrophy. Nat Med. 2019 Dec;25(12):1905-1915. doi: 10.1038/s41591-019-0669-y. Epub 2019 Dec 2. PMID 31792454
- [Derived] Tan L, Zschuntzsch J, Meyer S, Stobbe A, Bruex H, Regensburger AP, Classen M, Alves F, Jungert J, Rother U, Li Y, Danko V, Lang W, Turk M, Schmidt S, Vorgerd M, Schlaffke L, Woelfle J, Hahn A, Mensch A, Winterholler M, Trollmann R, Heiss R, Wagner AL, Raming R, Knieling F. Non-invasive optoacoustic imaging of glycogen-storage and muscle degeneration in late-onset Pompe disease. Nat Commun. 2024 Sep 8;15(1):7843. doi: 10.1038/s41467-024-52143-6. PMID 39245687
- See also: Publication of the clinical study — https://www.nature.com/articles/s41467-024-52143-6

DOCUMENTS (1):
  • Study Protocol (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05083806/Prot_000.pdf